CLINICAL TRIAL: NCT01857583
Title: Phase III Clinical Study of DU-176b (Venous Thromboembolism): Japanese, Multicenter, Open-label Study of DU-176b in Patients With Severe Renal Impairment (SRI) Undergoing Orthopedic Surgery of the Lower Limbs
Brief Title: Safety and Pharmacokinetics Study of DU-176b Administered to Patients With Severe Renal Impairment Undergoing Orthopedic Surgery of The Lower Limbs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DU176b-B-J306
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2015-02

CONDITIONS: Venous Thromboembolism
Keywords: anticoagulant; DU-176b; edoxaban; factor Xa; oral; orthopedic surgery of lower limbs; severe renal impairment
MeSH Terms: conditions — Venous Thromboembolism; Renal Insufficiency | interventions — edoxaban; Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SRI 15mg (15 mL/min ≤ CLCR < 20mL/min) (Experimental): Severe Renal Impairment group orally administered 15mg DU-176b once daily for 14 days.
  Interventions: Drug: 15mg DU-176b
- MiRI 30mg (50 mL/min ≤ CLCR ≤ 80mL/min) (Experimental): Mild Renal Impairment group orally administered 30mg DU-176b once daily for 14 days.
  Interventions: Drug: 30mg DU-176b
- Fondaparinux (20 mL/min ≤ CLCR < 30mL/min) (Active Comparator): Fondaparinux subcutaneously administered at a dose of 1.5mg once daily for 14 days.
  Interventions: Drug: Fondaparinux
- SRI 15mg (20 mL/min ≤ CLCR < 30mL/min) (Experimental): Severe Renal Impairment group orally administered 15mg DU-176b once daily for 14 days.
  Interventions: Drug: 15mg DU-176b

INTERVENTIONS:
Drug: 15mg DU-176b
  Other Names: edoxaban
  Arms: SRI 15mg (15 mL/min ≤ CLCR < 20mL/min); SRI 15mg (20 mL/min ≤ CLCR < 30mL/min)
Drug: 30mg DU-176b
  Other Names: edoxaban
  Arms: MiRI 30mg (50 mL/min ≤ CLCR ≤ 80mL/min)
Drug: Fondaparinux
  Arms: Fondaparinux (20 mL/min ≤ CLCR < 30mL/min)

SUMMARY:
To assess the safety and pharmacokinetics of DU-176b administered to patients with severe renal impairment undergoing orthopedic surgery of the lower limbs, compared with DU-176b administered to patients with mild renal impairment (MiRI) undergoing orthopedic surgery of the lower limbs.

For reference, the safety of DU-176b in patients with SRI undergoing orthopedic surgery of the lower limbs will be compared with that of fondaparinux.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SRI or MiRI undergoing orthopedic surgery of the lower limbs

Exclusion Criteria:

* Patients who are on hemodialysis or are scheduled to undergo hemodialysis during the study period
* Patients who are at a significantly high risk for bleeding or thromboembolism
* Patients who are receiving another antithrombotic therapy and are unable to suspend the therapy
* Patients who have evidence of hepatic function test abnormalities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Fuji, VP, Principal Investigator — Osaka Koseinenkin Hospital
Locations (1):
- Toyooka Chuo Hospital, Asahikawa, Hokkaido Prefecture, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Fuji T, Fujita S, Kawai Y, Abe Y, Kimura T, Fukuzawa M, Abe K, Tachibana S. A randomized, open-label trial of edoxaban in Japanese patients with severe renal impairment undergoing lower-limb orthopedic surgery. Thromb J. 2015 Jan 30;13(1):6. doi: 10.1186/s12959-014-0034-9. eCollection 2015. PMID 25653574

RESULTS

PARTICIPANT FLOW:
Groups:
- MiRI 30mg DU176b (50 mL/Min ≤ CLCR ≤ 80mL/Min): Mild Renal Impairment group orally administered 30mg DU176b once daily for 14 days.
  (50 mL/min ≤ CLCR ≤ 80 mL/min) 30mg DU-176b
- SRI 15mg DU176b (15 mL/Min ≤ CLCR < 20 mL/Min): Severe Renal Impairment group orally administered 15mg DU-176b once daily for 14 days.
  (15 mL/min ≤ CLCR < 20 mL/min) 15mg DU-176b
- SRI 15mg DU176b (20 mL/Min ≤ CLCR < 30 mL/Min): Severe Renal Impairment group orally administered 15mg DU176b once daily for 14 days.
  (20 mL/min ≤ CLCR < 30 mL/min) 15mg DU-176b
- Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min): Fondaparinux subcutaneously administered at a dose of 1.5mg once daily for 14 days.
  (20 mL/min ≤ CLCR < 30mL/min) Fondaparinux
Period: Overall Study
Arm/Group | MiRI 30mg DU176b (50 mL/Min ≤ CLCR ≤ 80mL/Min) | SRI 15mg DU176b (15 mL/Min ≤ CLCR < 20 mL/Min) | SRI 15mg DU176b (20 mL/Min ≤ CLCR < 30 mL/Min) | Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min)
Started | 30 | 7 | 22 | 21
Safety Analysis Population | 30 | 7 | 22 | 20
Completed | 29 | 6 | 19 | 17
Not Completed | 1 | 1 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Death | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The number of baseline participants reflects the safety analysis population.
Groups:
- MiRI 30mg DU176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min): Mild Renal Impairment group orally administered 30mg DU176b once daily for 14 days.
  (50 mL/min ≤ CLCR ≤ 80 mL/min) 30mg DU-176b
- Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min): Fondaparinux subcutaneously administered at a dose of 1.5mg once daily for 14 days.
  (20 mL/min ≤ CLCR < 30mL/min)
- Total: Total of all reporting groups
Arm/Group | MiRI 30mg DU176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min) | SRI 15mg DU176b (15 mL/Min ≤ CLCR < 20 mL/Min) | SRI 15mg DU176b (20 mL/Min ≤ CLCR < 30 mL/Min) | Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min) | Total
Number analyzed (Participants) | 30 | 7 | 22 | 20 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.1 (6.46) | 91.7 (7.06) | 86.5 (4.31) | 85.7 (8.91) | 83.5 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 6 | 19 | 20 | 72
  Male | 3 | 1 | 3 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 30 | 7 | 22 | 20 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Any Adjudicated Bleeding Events
Description: Incidence of any adjudicated bleeding events (including major bleeding, clinically relevant non-major bleeding, and minor bleeding).
Time Frame: 14 days
Population: The safety analysis set was defined as all subjects who were enrolled in the study, except for those who had significant GCP violations, who had not received the study drug, or who had no safety data after the start of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of subjects with bleeds
Groups:
- MiRI 30mg DU 176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min): Mild Renal Impairment group orally administered 30mg DU176b once daily for 14 days.
  (50 mL/min ≤ CLCR ≤ 80 mL/min) 30mg DU-176b
- SRI 15mg DU 176b (15 mL/Min ≤ CLCR < 20 mL/Min): Severe Renal Impairment group orally administered 15mg DU-176b once daily for 14 days.
  (15 mL/min ≤ CLCR < 20 mL/min) 15mg DU-176b
- SRI 15mg DU 176b (20 mL/Min ≤ CLCR < 30 mL/Min): Severe Renal Impairment group orally administered 15mg DU176b once daily for 14 days.
  (20 mL/min ≤ CLCR < 30 mL/min) 15mg DU-176b
Arm/Group | MiRI 30mg DU 176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min) | SRI 15mg DU 176b (15 mL/Min ≤ CLCR < 20 mL/Min) | SRI 15mg DU 176b (20 mL/Min ≤ CLCR < 30 mL/Min) | Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min)
Number analyzed (Participants) | 30 | 7 | 22 | 20
percentage of subjects with bleeds | 33.3 [19.2 to 51.2] | 14.3 [2.6 to 51.3] | 22.7 [10.1 to 43.4] | 40.0 [21.9 to 61.3]
Statistical Analysis 1: Comparison: MiRI 30mg DU 176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min) vs SRI 15mg DU 176b (15 mL/Min ≤ CLCR < 20 mL/Min) vs SRI 15mg DU 176b (20 mL/Min ≤ CLCR < 30 mL/Min); Test type: Superiority or Other; ANCOVA; Cox Proportional Hazard = 12.6, 95% CI 2-sided [-10.0 to 33.6]
Statistical Analysis 2: Comparison: SRI 15mg DU 176b (20 mL/Min ≤ CLCR < 30 mL/Min) vs Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min); Test type: Superiority or Other; ANCOVA; Cox Proportional Hazard = 17.3, 95% CI 2-sided [-10.2 to 42.1]

2. Primary Outcome: Incidence of Adverse Events
Time Frame: 1 month
Reporting Status: Not Posted

3. Primary Outcome: Incidence of Adverse Drug Reactions
Time Frame: 1 month
Reporting Status: Not Posted

4. Primary Outcome: Plasma Concentration of DU-176b
Time Frame: 14 days
Reporting Status: Not Posted

5. Primary Outcome: Plasma Concentration of D21-2393
Time Frame: 14 days
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Adjudicated Thromboembolic Events
Description: Incidence of adjudicated thromboembolic events (symptomatic Deep Vein Thrombosis (DVT), symptomatic Pulmonary Thromboembolism (PTE), Venous Thromboembolism (VTE) related deaths).
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min): Fondaparinux subcutaneously administered at a dose of 1.5mg once daily for 14 days.
  Fondaparinux (20 mL/min ≤ CLCR < 30mL/min)
Arm/Group | MiRI 30mg DU 176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min) | SRI 15mg DU 176b (15 mL/Min ≤ CLCR < 20 mL/Min) | SRI 15mg DU 176b (20 mL/Min ≤ CLCR < 30 mL/Min) | Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min)
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/7 | 2/22 | 3/20
Other Adverse Events (participants affected / at risk) | 22/30 | 6/7 | 12/22 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiRI 30mg DU 176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min) (N=30) | SRI 15mg DU 176b (15 mL/Min ≤ CLCR < 20 mL/Min) (N=7) | SRI 15mg DU 176b (20 mL/Min ≤ CLCR < 30 mL/Min) (N=22) | Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min) (N=20)
cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiRI 30mg DU 176b (50 mL/Min ≤ CLCR ≤ 80 mL/Min) (N=30) | SRI 15mg DU 176b (15 mL/Min ≤ CLCR < 20 mL/Min) (N=7) | SRI 15mg DU 176b (20 mL/Min ≤ CLCR < 30 mL/Min) (N=22) | Fondaparinux (20 mL/Min ≤ CLCR < 30mL/Min) (N=20)
cystitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 6 (9) | 0 (0) | 1 (2) | 3 (4)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pubic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 2 (2) | 4 (4) | 0 (0)
Blood urine present (Investigations) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Red blood cells urine positive (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.